CLINICAL TRIAL: NCT01625663
Title: Heart and Skeletal Muscle Metabolism, Energetics and Function in Barth Syndrome
Brief Title: Heart and Muscle Metabolism in Barth Syndrome
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105474
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Barth Syndrome
Keywords: barth syndrome; heart failure; mitochondria; metabolism; amino acid
MeSH Terms: conditions — Barth Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, skin biopsy, breath, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Barth syndrome: Children (8-17 yrs) and adults (18-35 yrs)
- Controls: Children (8-15 yrs) and adults (18-35 yrs)

SUMMARY:
Barth syndrome (BTHS) is an X-linked disorder caused by abnormal cardiolipin metabolism and is characterized by skeletal and cardiomyopathy and high mortality rates. Through clinical metabolism and imaging studies and pluripotent stem cell induction and molecular techniques on skin biopsy samples, this project will produce novel translational information regarding the pathogenesis of BTHS, reveal potential targets for interventions and provide unique data regarding nutrient metabolism and abnormal cardiolipin and mitochondrial function. This project has the potential to provide information that could significantly improve morbidity and mortality in children and young adults with BTHS and may have relevance to other non-BTHS related conditions such as aging and adult heart failure.

DETAILED DESCRIPTION:
Barth syndrome (BTHS) is an X-linked disorder characterized by abnormal cardiolipin metabolism, mitochondrial dysfunction, muscle wasting and heart failure. BTHS is a particularly significant disease as it is often fatal in childhood and there are no approved therapies for BTHS other than the standard treatment of heart failure. Therefore novel areas of research and platforms in which to test new therapies are highly needed. Through state-of-the-art and innovative methodologies, this project will focus on the novel role of skeletal muscle and heart nutrient (glucose, fatty acid, and amino acid) metabolism in the pathogenesis of BTHS. Phenotypic information regarding skeletal muscle and heart nutrient metabolism in BTHS and how it may relate to energy production and function of these organs is lacking and is significant as this may advance our understanding of the underlying pathogenesis of BTHS. With this understanding, safe and efficacious therapies can be targeted for BTHS. The investigators' overall hypothesis is that impaired fatty acid metabolism in skeletal muscle and the heart produces a fuel deficit in these organs leading to impaired energy production, exercise intolerance and heart failure. Further, as a consequence of impaired fatty acid metabolism in skeletal muscle and the heart, protein breakdown (wasting) in skeletal muscle and the heart occurs to provide amino acids as compensation for this inadequate fatty acid energy supply, thereby worsening heart and skeletal muscle function in BTHS. The investigators' aims to address this hypothesis in 30 young adults and children with BTHS and 30 healthy, age, puberty stage and activity level matched controls ages 8-35 years are:

1) To characterize skeletal muscle and heart nutrient metabolism and 2) To examine the relationship between skeletal muscle and heart nutrient metabolism, energy production and function (exercise tolerance and heart function). As an exploratory aim, we will examine mechanistic molecular pathways of nutrient metabolism; specifically protein breakdown, mitochondrial function and fatty acid metabolism, in human myocytes derived from inducible pluripotent stem cells (from skin fibroblasts) obtained from adults and children with BTHS and from adult controls. Skeletal muscle nutrient metabolism will be quantified by stable-isotope tracer methodology and mass spectrometry, heart nutrient metabolism using radio-isotope tracer methodology and PET imaging, skeletal muscle and heart energy production using magnetic resonance spectroscopy, skeletal muscle function by graded exercise testing and indirect calorimetry, heart function by echocardiography, and myocyte nutrient pathway mechanism examination by pluripotent stem cell induction and protein and RNA expression analyses.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of BTHS or healthy control
2. age 8-35 years
3. sedentary (physically active less than 2x/wk)
4. stable on medications for ≥ 3 months including ß-blockers, ACE inhibitors, digoxin
5. lives in North America, the UK, Europe, South Africa or other locations feasible for travel to the US

Exclusion Criteria:

1. current unstable heart disease
2. diabetes or other known concurrent disease that may affect nutrient metabolism

Ages: 8 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adults ages 8-35 yrs with Barth syndrome and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Whole-body fatty acid oxidation rate | baseline
  Whole-body fatty acid oxidation rate will be measured by 13C-labeled fatty acid stable isotope tracer infusion and mass spectrometry

SECONDARY OUTCOMES:
whole-body amino acid oxidation rate | baseline
  whole-body amino acid oxidation rate will be measured by 13C leucine stable isotope tracer infusion and mass spectrometry
cardiac energetics | baseline
  cardiac energetics will be measured by 31P magnetic resonance spectroscopy of the heart
skeletal muscle energetics | baseline
  skeletal muscle energetics will be measured by 31P magnetic resonance spectroscopy
Myocardial fatty acid oxidation rate | baseline
  Myocardial fatty acid oxidation rate will be measured by radio-isotope tracer infusion and PET imaging
left ventricular systolic strain | baseline
  Left ventricular systolic strain will be measured by tissue Doppler echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: William T Cade, PT, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Result] Cade WT, Bohnert KL, Peterson LR, Patterson BW, Bittel AJ, Okunade AL, de las Fuentes L, Steger-May K, Bashir A, Schweitzer GG, Chacko SK, Wanders RJ, Pacak CA, Byrne BJ, Reeds DN. Blunted fat oxidation upon submaximal exercise is partially compensated by enhanced glucose metabolism in children, adolescents, and young adults with Barth syndrome. J Inherit Metab Dis. 2019 May;42(3):480-493. doi: 10.1002/jimd.12094. Epub 2019 Apr 11. PMID 30924938
- [Result] Bashir A, Bohnert KL, Reeds DN, Peterson LR, Bittel AJ, de las Fuentes L, Pacak CA, Byrne BJ, Cade WT. Impaired cardiac and skeletal muscle bioenergetics in children, adolescents, and young adults with Barth syndrome. Physiol Rep. 2017 Feb;5(3):e13130. doi: 10.14814/phy2.13130. PMID 28196853
- [Derived] Cade WT, Laforest R, Bohnert KL, Reeds DN, Bittel AJ, de las Fuentes L, Bashir A, Woodard PK, Pacak CA, Byrne BJ, Gropler RJ, Peterson LR. Myocardial glucose and fatty acid metabolism is altered and associated with lower cardiac function in young adults with Barth syndrome. J Nucl Cardiol. 2021 Aug;28(4):1649-1659. doi: 10.1007/s12350-019-01933-3. Epub 2019 Nov 8. PMID 31705425